CLINICAL TRIAL: NCT06020703
Title: Healthy Microbiome, Healthy Mind: Using Gut-brain Axis for Improving Psychocognitive Health Outcomes of Critical Illness Survivors
Brief Title: A Study of Healthy Microbiome, Healthy Mind
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Lioudmila Karnatovskaia, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-005057
Record Dates: First submitted 2023-08-23; First posted 2023-09-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Critical Illness; COVID-19; PICS; Cognitive Impairment; Mental Health Impairment; Weakness, Muscle; Dysbiosis
MeSH Terms: conditions — Critical Illness; COVID-19; Cognitive Dysfunction; Muscle Weakness; Dysbiosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermented Foods Diet (Experimental): Subjects will incorporate fermented food into their diet.
  Interventions: Behavioral: Fermented Food Diet
- Normal Diet (No Intervention): Subjects will continue their regular diet.

INTERVENTIONS:
Behavioral: Fermented Food Diet — Subjects will incorporate 1 serving of fermented food a day and increase to 6 more each day as tolerated for 4 weeks. After the initial 4 weeks, subjects will eat 6 or more servings of fermented foods each day for 8 weeks.
  Arms: Fermented Foods Diet

SUMMARY:
Researchers are doing this study to find out if a high fermented food diet is tolerable, and if it will help improve quality of life after surviving a critical illness, including severe COVID-19, by promoting gut health recovery and decreasing gut inflammation.

DETAILED DESCRIPTION:
Critical illness, including severe COVID, often lead to long term cognitive and mental health complications. Current non-pharmacological interventions, including ABCDEF bundle, are of limited efficacy. The largest psychological intervention trial to date also demonstrated no beneficial effect. These impairments may persist for years and are associated with chronic pain, impaired physical functioning, decreased quality of life, increased use of psychotropic medications, opioid abuse, self-harm, and increased acute care service utilization. Half of previously employed critical illness survivors, including those with long COVID, are not able to return to work a year later resulting in loss of insurance and difficulty in seeking professional help.

Increasing recognition that the nervous system and the gastrointestinal tract are communicating through a bidirectional network of signaling pathways, collectively known as the gut-brain-axis, resulted in emergence of a novel discipline of "nutritional psychiatry" advocating that diet and nutrition may be central determinants of both physical and mental health. In the outpatient setting, fiber rich Mediterranean style diet has been linked to improvements in cognitive and mood symptoms possibly via its known anti-inflammatory effect whereby diets high in sugars and refined grains with high inflammatory potential have been linked to the development of depression.

Critical illness and associated interventions lead to the loss of normal gut bacteria, allowing overgrowth of disease-promoting pathogenic bacteria resulting in severe dysbiosis. During dysbiosis, gut-brain pathways are dysregulated resulting in neuroinflammation, anxiety and depressive-like behaviors as well as cognitive impairment. Dysbiosis can persist months after the resolution of critical illness. Restoration of healthy microbiome may thus be key to facilitating psychiatric and cognitive recovery after critical illness.

Can the Mediterranean diet be used to restore microbiome diversity in this population? Perhaps not right away, as critical illness survivors have significant decrease in fiber degrading bacterial organisms. Others demonstrated that high-fiber diet alone does not result in increased microbial community diversity. What about probiotics? In patients with antibiotics-associated dysbiosis, probiotics induced a persistently incomplete indigenous stool microbiome recovery. How can microbiome diversity be restored? Fermented foods may be the most promising approach. Consumption of fermented milk facilitated restoration of gut homeostasis in patients with irritable bowel syndrome and increased their "feeling good" scores. Other human intervention studies using fermented tea, sauerkraut, fermented plant extract, kimchi, and fermented soybean milk reported increased presence of bacteria in the gut known for their health promoting properties. Consumption of fermented foods was associated with positive modulation in brain activity and fewer symptoms of social anxiety. A 10-week high fermented food diet intervention demonstrated increased microbiota diversity and decreased inflammatory markers among healthy volunteers. Can it be applied to survivors of critical illness including COVID to help them recover from dysbiosis and inflammation, and improve their mental health and other outcomes?

Specific Aim #1: to evaluate feasibility of high fermented food diet among critical illness survivors and its effect on microbiome diversity Hypothesis 1a: critical illness survivors will tolerate high fermented food diet Hypothesis 1b: high fermented food diet will increase microbiome diversity in critical illness survivors.

Specific Aim #2: to evaluate the effect of high fermented food diet on immune system performance and recovery, mental health, cognition, and quality of life of critical illness survivors.

Hypothesis 2a: high fermented food diet will improve immune system performance among critical illness survivors.

Hypothesis 2b: critical illness survivors treated with fermented food diet for 3 months will have a reduction in symptoms of anxiety, depression and acute stress/PTSD Hypothesis 2c: critical illness survivors treated with fermented food diet for 3 months will have improvement in cognition.

Hypothesis 2c: critical illness survivors treated with fermented food diet for 3 months will have improvement in quality of life.

ELIGIBILITY:
Inclusion Criteria:

- patients who have survived critical illness, including severe COVID, and are at risk for mental health morbidity/long COVID (spent >48 hours in the ICU or had COVID requiring ICU stay) who have a smartphone, are enrolled into the Mayo PICS clinic, and have at least one PICS-related impairment. Cognitive impairment, if present, has to be in the mild range to ensure patient can provide consent and follow study instructions

Exclusion Criteria:

- History of dementia, mental retardation, psychotic disorders such as schizophrenia, patients not expected to survive the hospital stay or non-English speaking, participants not able to tolerate foods by mouth or those with potential contraindications to such diet (chronically immunosuppressed including organ transplant recipients; those with neutropenia or currently undergoing chemotherapy, those taking Monoamine oxidase inhibitors).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of high fermented food diet among critical illness survivors | 12 weeks
  20 critical illness survivors assigned to the intervention arm will tolerate high fermented food diet on 75% of the study days or more
gut microbiome diversity | Baseline, 12 weeks
  assessed using Shannon index

SECONDARY OUTCOMES:
Change in inflammatory cytokines | Baseline, 12 weeks
  Targeted analyses will be performed to compare the values of inflammatory markers such as tumor necrosis factor-alpha, interleukin-2, interleukin-2 soluble receptor, interleukin-4, interleukin-5, interleukin-6, interleukin-8, interleukin-10, interleukin-12 interleukin-13, interleukin-17, interferon-gamma and interferon-1beta. All marker levels are measured in pg/ml.
Symptoms of anxiety and depression | Baseline, 12 weeks
  Measured using the self-reported Hospital Anxiety and Depression Scale (HADS). Total questions: 14. Anxiety 7, Depression 7. Each item is rated on a 4-point scale from 0 "absence" to 3 "extreme presence". Total score is 21 per subscale: 0 - 7: Normal levels of anxiety/depression; 8-10: Borderline abnormal; > 11: Abnormal
Cognitive Assessment | Baseline, 12 weeks
  Measured using the Montreal Cognitive Assessment (MoCA-BLIND). Total questions:13. Memory 3 Attention 4 Language 3 Abstraction 2 Orientation 1. Subscores for each of the 5 sections are calculated. The total score is summed from the subscores, with a maximum score of 22. A score equal > 18 is considered normal cognition
Self-Reported quality of life | Baseline, 12 weeks
  Measured using the self-reported EuroQol-5D-3L questionnaire. Total questions: 6. Mobility: 1, Self-Care: 1, Usual Activities: 1, Pain/discomfort: 1, Anxiety/depression: 1, Health State - Visual Analog Scale: 1. 3L - 3 levels of severity: no problems, some problems, extreme problems. The visual analog scale ranges from 0 to 100 with higher scores reflecting better perceived current health-related quality of life state.
symptoms of acute stress/PTSD | Baseline, 12 weeks
  Measured using Impact of Events-revised (IES-r). Total questions: 22. Intrusion 7, Avoidance 8, Hyperarousal 7. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Total scores are summed with higher scores indicating greater distress with regards to a specific event.
  Orientation 1

CONTACTS AND LOCATIONS:
Overall Officials: Lioudmila Karnatovskaia, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No